CLINICAL TRIAL: NCT02472587
Title: Assessing Chronic Pain Conditions in General Population
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Other Study IDs: PelvicPain
Record Dates: First submitted 2015-06-07; First posted 2015-06-16 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Pelvic Pain
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pap test: Women attending our institute in order to do Pap test
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
The purpose of this study is to determine the percentage of women, among those attending our institute in order to do Pap test, suffering of chronic pelvic pain. To such purpose the patients will be submitted to questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age

Exclusion Criteria:

* unwilling or unable to give consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women attending our institute in order to do Pap test
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Chronic pelvic pain Questionnaire | 5 years